CLINICAL TRIAL: NCT00001080
Title: Effect of Vaccination on Turnover of Lamivudine (3TC) Sensitive and Resistant Virus Populations in HIV-1-Infected Individuals
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: as of 4/23/97
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 340; 11311 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Lymphocyte Transformation; HIV-1; Drug Resistance, Microbial; CD4-Positive T-Lymphocytes; Lamivudine; Influenza Vaccine; RNA, Viral; Bacterial Vaccines; Anti-HIV Agents; Pneumonia, Pneumococcal; Viral Load
MeSH Terms: conditions — HIV Infections; Influenza, Human; Pneumonia, Pneumococcal | interventions — Influenza Vaccines; Pneumococcal Vaccines; Lamivudine

INTERVENTIONS:
Biological: Influenza Virus Vaccine
Biological: Pneumococcal Vaccine, Polyvalent (23-valent)
Drug: Lamivudine

SUMMARY:
To ascertain whether the origin of plasma HIV-1-RNA following T cell activation represents the activation of latently infected cells or an increase in cells permissive for replacing viral mutants.

The mechanism by which immune stimulation increases circulating levels of HIV-1 is not known. In particular, it is uncertain whether the transient increase in plasma HIV-1 RNA is due to enhanced replication of an actively replicating pool of HIV-1, or is due instead to activation of proviral sequences in previously resting CD4+ cells. One approach to discriminate these alternatives is a "molecular pulse-chase" experiment. In this approach, drug resistant mutants would be selected by administration of Lamivudine (3TC).

DETAILED DESCRIPTION:
The mechanism by which immune stimulation increases circulating levels of HIV-1 is not known. In particular, it is uncertain whether the transient increase in plasma HIV-1 RNA is due to enhanced replication of an actively replicating pool of HIV-1, or is due instead to activation of proviral sequences in previously resting CD4+ cells. One approach to discriminate these alternatives is a "molecular pulse-chase" experiment. In this approach, drug resistant mutants would be selected by administration of Lamivudine (3TC).

Twenty subjects without prior 3TC experience will be treated with 3TC for 2 weeks. On day 14, half of the subjects will receive immunization with both the influenza and pneumococcal vaccine. 3TC will be discontinued at this time. Patients will be followed for 4 weeks after the immunization.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy, provided the patient has been on the same dose and drugs for 60 days prior to study entry.

Patients must have:

* Documented HIV infection.
* CD4 lymphocyte count of > 300 cells/mm3.
* One plasma HIV-1 RNA level between >= 20,000 and < 120,000 copies/ml.

Prior Medication:

Allowed:

* Stable antiretroviral therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Presence of an AIDS defining opportunistic infection, including Kaposi's sarcoma.
* Allergy to influenza or pneumococcal vaccine or their components; to egg or egg products.
* Unexplained temperature >= 38.5 degrees C for 7 consecutive days within the 30 days prior to study entry.
* Concurrent participation in other experimental therapies.

Concurrent Medication:

Excluded:

* Systemic chemotherapy.
* Steroids.
* Corticosteroids.
* Vaccinations.
* Any new antiretroviral agents that the patient was not taking at the time of study entry and not prescribed by the study.
* Colony stimulating factors including G-CSF or rEPO.
* Immune modulators/immune based therapies.

Concurrent Treatment:

Excluded:

* Radiation therapy.
* Transfusion dependent patients.

Patients with any of the following prior conditions are excluded:

* History of an AIDS defining opportunistic infection, including Kaposi's sarcoma (except limited cutaneous diseases [< 5 lesions]).
* History of acute or chronic pancreatitis.

Prior Medication:

Excluded:

* Prior treatment with 3TC.

Excluded within 30 days of study entry:

* Treatment with immune modulators.
* Acute or chronic therapy for recognized infections (eg, influenza, HSV, VZV).

Excluded within 1 year of study entry:

Treatment with an influenza and/or pneumonia vaccine

[AS PER AMENDMENT 1/23/97:

* influenza vaccine only].

[AS PER AMENDMENT 1/23/97:

* Excluded within 3 years of study entry:
* Pneumonia vaccine.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuritzkes D, Study Chair; Richman D, Study Chair; Havlir D, Study Chair